CLINICAL TRIAL: NCT06094166
Title: Quantitative Magnetic Resonance Imaging Parameters as Predictors of Outcome for Non-Myelopathic Degenerative Cervical Cord Compression: A Longitudinal Study
Brief Title: Quantitative MR Parameters in Non-myelopathic Degenerative Cervical Spinal Cord Compression: a Longitudinal Study.
Acronym: NOLOST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Masaryk University (Other)
Collaborators: Palacky University (Other)
Responsible Party: Principal Investigator, Tomáš Horák, prof. MUDr. Josef Bednarik, CSc., FCMA, FEAN, Masaryk University
Other Study IDs: 66138
Record Dates: First submitted 2023-09-12; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Degenerative Cervical Spinal Myelopathy; Cervical Spinal Cord Compression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NMDCC: non-myelopathic cervical spinal cord compression
  Interventions: Diagnostic Test: MRI
- healthy controls: subjects with no MR signs of cervical spinal cord compression
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Quantitative imaging MR parameters

SUMMARY:
Quantitative Magnetic Resonance Imaging Parameters as Predictors of Outcome for Non-Myelopathic Degenerative Cervical Cord Compression: A Longitudinal Study

DETAILED DESCRIPTION:
The study uses semi-automated detection of anatomical metrics (morphometric parameters) and DCC with Spinal Cord Toolbox (SCT). This method have been proven more reliable than expert's manual rating, the introduction of the automated method will be utilized in the future multi-centre and longitudinal studies. Routine anatomical morphometric parameters such as compressive ratio (CR) and cross-sectional area (CSA) will be acquired along with microstructural and metabolic metrics obtained with validated dMRI and MRS methods, remote cervical cord atrophy from voxel-based MRI volumetry, T2* white matter/gray matter (WM/GM) signal-intensity ratio, and also metrics obtained with novel Intravoxel Incoherent Motion (IVIM) method will predict progression of NMDCC into symptomatic DCM. "Natural course" (i.e., speed of progression) of the severity of DCC assessed with anatomical and advanced MRI/MRS metrics is not known but may play a role in the progression from NMDCC to symptomatic DCM. Aims of this project are: To determine independent predictors of unfavourable outcome - progression into symptomatic degenerative cervical myelopathy (DCM) - among quantitative MRI parameters and compare them with already defined clinical and electrophysiological predictors. To evaluate the "natural course" of MRI descriptors of compression and its severity, and the correlation between progression and development of symptomatic DCM. To implement automated detection of cervical cord compression using Spinal Cord Toolbox based on automatically computed morphometric parameters.

ELIGIBILITY:
Inclusion Criteria:

Subject with no contraindication to MR examination. Clinically asymptomatic cervical spinal cord compression or subjects with no spinal cord compression.

Exclusion Criteria:

* A subject will be excluded if he/she has a contraindication to MR scanning implanted metal clips or wires of the type which may concentrate radiofrequency fields or cause tissue damage from twisting in a magnetic field.
* Pregnancy
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls and patients with non-myelopathic cervical spinal cord compression (NMDC)
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Anatomical MRI metrics | 45 minutes
  compressive ratio (CR)
Anatomical MRI metrics | 45 minutes
  cross-sectional area (CSA)
dMRI: signs of microstructural myelopathy | 45 minutes
  fractional anisotropy
MRS: signs of metabolic myelopathy (above the level of compression) | 45 minutes
  Myo-ins/NAA ratio
Voxel-based MRI volumetry (remote spinal cord atrophy above the compression level) | 45 minutes
  remote cervical cord atrophy

SECONDARY OUTCOMES:
IVIM and T2*WM/GM signal-intensity ratio | 45 minutes
  Intravoxel incoherent motion detection

CONTACTS AND LOCATIONS:
Overall Officials: Josef Bednarik, Prof. MD., Principal Investigator — Masaryk University
Locations (1):
- Faculty of Medicine, Masaryk University, Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided